CLINICAL TRIAL: NCT01383382
Title: Transforming PCI Informed Consent Into an Evidence-based Decision-making Tool
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Washington University School of Medicine (Other); Baylor Research Institute (Other); Baystate Medical Center (Other); Henry Ford Health System (Other); Kaiser Permanente (Other); Prairie Education and Research Cooperative (Industry)
Responsible Party: John A. Spertus, MD, MPH, Saint Luke's Hospital of Kansas City
Other Study IDs: R01HL096624 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2011-06

CONDITIONS: Non-emergent Percutaneous Coronary Intervention (PCI)
Keywords: Heart Diseases; Cardiovascular Diseases; Acute Myocardial Infarction; Decision Making; Percutaneous Coronary Intervention; Informed Consent; Quality of Care
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Using individualized patient estimates of procedural risks and benefits, this project will transform the process of informed consent for coronary angioplasty into a dynamic educational tool for patients and physicians and is a direct response to the Institute of Medicine's call for a more evidence-based, efficient, patient-centered healthcare system. It is hypothesized that patients will develop a greater understanding of their individual risks and benefits from PCI, will be empowered to more actively engage in shared decision-making, as well as have improved awareness of their responsibility to adhere to dual anti-platelet therapy if treated with a drug eluting stent (risks for target vessel revascularization with bare metal and drug eluting stents are also provided in the new consent form). It is also anticipated that physicians, in turn, will use these individualized estimates to better discriminate between risks and benefits among different bleeding avoidance therapies so as to improve the safety and cost-effectiveness of PCI.

DETAILED DESCRIPTION:
This study will test the impact of a new mechanism for eliciting informed consent from patients undergoing percutaneous coronary intervention (PCI) on 1) patients' comprehension of procedural risks/benefits and participation in shared decision-making; and 2) upon clinicians' use of effective strategies to minimize the risk of bleeding at the time of PCI. To facilitate these goals, we will prospectively provide each patients' risks for bleeding at the time that the informed consent document is generated. This will be accomplished by transforming the infrastructure of the informed consent process at participating study centers using a novel, web-based system - the Personalized Risk Information Services Manager (PRISM) - to generate individualized consent forms with estimates of risks and outcomes using validated multivariable models from the American College of Cardiology's NCDR. The goals of this study are to 1) identify barriers in implementing individualized consent forms in clinical care and to test whether this novel consent process 2) improves the quality of the informed consent process, 3) supports the more rational use of Bleeding Avoidance Therapies (BATs), 4) reduces bleeding events after PCI, and 5) supports a more cost-effective PCI procedure. This will be done using a pre-post design at 6 enrolling hospitals and comparing changes in practice with contemporaneous controls matched from the broader NCDR Cath/PCI registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a PCI in a participating institution

Exclusion Criteria:

* Previously enrolled in the PRISM
* Does not speak English or Spanish
* Dementia
* Too ill to interview
* Current prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac patients undergoing a non-emergent percutaneous coronary intervention (PCI) procedure for their heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 1399 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Spertus, MD, MPH, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri
Locations (7):
- United States (7):
  - Kaiser Permanente, Oakland, California
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes-Jewish Hospital/Washington University School of Medicine, St Louis, Missouri
  - Baylor Research Institute, Plano, Texas

REFERENCES:
- [Derived] Spertus JA, Decker C, Gialde E, Jones PG, McNulty EJ, Bach R, Chhatriwalla AK. Precision medicine to improve use of bleeding avoidance strategies and reduce bleeding in patients undergoing percutaneous coronary intervention: prospective cohort study before and after implementation of personalized bleeding risks. BMJ. 2015 Mar 24;350:h1302. doi: 10.1136/bmj.h1302. PMID 25805158
- [Derived] Spertus JA, Bach R, Bethea C, Chhatriwalla A, Curtis JP, Gialde E, Guerrero M, Gosch K, Jones PG, Kugelmass A, Leonard BM, McNulty EJ, Shelton M, Ting HH, Decker C. Improving the process of informed consent for percutaneous coronary intervention: patient outcomes from the Patient Risk Information Services Manager (ePRISM) study. Am Heart J. 2015 Feb;169(2):234-241.e1. doi: 10.1016/j.ahj.2014.11.008. Epub 2014 Nov 15. PMID 25641532
- [Derived] Safley DM, Grantham JA, Hatch J, Jones PG, Spertus JA. Quality of life benefits of percutaneous coronary intervention for chronic occlusions. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):629-34. doi: 10.1002/ccd.25303. Epub 2013 Dec 19. PMID 24259445